CLINICAL TRIAL: NCT01117467
Title: Factors Affecting Medical Student Learning in Simulation Scenarios
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Principal Investigator, Imogen Davies, Clinical Lecturer, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 10/H0501/7
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Learning
Keywords: Simulation; Learning; Medical Students; Empathy; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Solo (Experimental): Students will perform their simulation scenario solo and receive feedback within the group
  Interventions: Other: Simulation scenario
- Paired (Experimental): Students will be paired with one of their peers for this simulation scenario
  Interventions: Other: Simulation scenario

INTERVENTIONS:
Other: Simulation scenario — Students performing their scenario will be paired, not solo
  Arms: Paired
Other: Simulation scenario — Students will perform their simulation scenario solo and receive feedback within the group
  Arms: Solo

SUMMARY:
Simulation is used to teach undergraduate and postgraduate healthcare professionals, however it is not known how best to use this resource. Using qualitative methods, this study aims to investigate how medical students learn during simulation scenarios and will compare students who are paired with peers with those who are solo during their scenarios. Video and audio data from simulations will be collected and analysed with anxiety and empathy questionnaire data and semi-structured interviews.

DETAILED DESCRIPTION:
Medical students attending a simulation day will either perform their simulation paired with another student from the group or solo. Video data from the scenario and audio data from the feedback session will be retained. One week later students will perform a second scenario and the feedback following this will be retained. Students will also have a semi-structured interview and complete anxiety and empathy questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* All final year medical students at the study university who are allocated to attend the anaesthesia special study module

Exclusion Criteria:

* Non-English speakers
* Visiting students who will be unable to complete the study
* Students who refuse to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Learning during simulation scenario as measured qualitatively | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Imogen Davies, MB BCh, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom